CLINICAL TRIAL: NCT03686488
Title: A Phase II Study of TAS 102 in Combination With Ramucirumab in Advanced, Refractory Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: TAS 102 in Combination With Ramucirumab in Advanced, Refractory Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19477
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — trifluridine tipiracil drug combination; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS 102 and Ramucirumab (Experimental): TAS 102 (Lonsurf) and Ramucirumab 10 MG/ML Intravenous Solution (CYRAMZA) administered concurrently.
  Interventions: Drug: TAS 102; Drug: Ramucirumab 10 MG/ML Intravenous Solution [CYRAMZA]

INTERVENTIONS:
Drug: TAS 102 — TAS 102 35 mg will be administered orally twice daily every 2 weeks.
  Other Names: Lonsurf
Drug: Ramucirumab 10 MG/ML Intravenous Solution [CYRAMZA] — Ramucirumab 8 milligrams/kilogram will be administered as a 60 minute intravenous (IV) infusion every 2 weeks.

SUMMARY:
The purpose of this study is to find out if the combination of TAS 102 and Ramucirumab is safe and effective in patients with advanced, refractory gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of gastric and GEJ adenocarcinoma.
* Measurable or non-measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Stage IV or recurrent disease is required. An irradiated lesion is considered evaluable only if it has shown enlargement since the completion of last radiation.
* Participants must have received and progressed with prior therapy. Prior therapy with ramucirumab is not allowed. Participants must have recovered from the toxic effects of the previous anti-cancer chemotherapy (with the exception of alopecia).
* Eastern Cooperative Oncology Group (ECOG) Performance score 0 or 1
* Estimated life expectancy > 3 months
* Adequate bone marrow, liver and renal function as assessed by the following: Hemoglobin > 8.0 g/dl, Absolute neutrophil count (ANC) > 1,000/mm3 independent of growth factor support, Platelet count > 100,000/mm3, Total bilirubin < 1.5 times upper limits of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, aspartate transaminase (AST), alanine transaminase (ALT) and Alkaline Phosphatase ≤2.5 times the ULN ( ≤5 x ULN for patients with liver involvement), Creatinine clearance ≥ 30 ml/min.
* Participants must not have had chemotherapy,major surgery, monoclonal antibody therapy or experimental therapy within the 28 days prior to the start of TAS 102 administration.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Participants (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form until at least 4 months for both females and males after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Participants must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.

Exclusion Criteria:

* Participants with active Central Nervous System (CNS) metastases are excluded. If CNS metastases are treated and participants are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment.
* Women who are pregnant or breast-feeding.
* Prior therapy with ramucirumab, bevacizumab, regorafenib or TAS 102.
* Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder 15 tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Uncontrolled hypertension (systolic BP >140 mm Hg or diastolic BP >90 mm Hg on repeated measurement despite optimal medical management)
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Persistent proteinuria ≥ Grade 3 on repeated measurement.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Participants with an arterial thrombotic or thromboembolic event within 12 months of informed consent.
* Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Clinically significant cardiovascular disease such as unstable angina, uncontrolled or symptomatic arrhythmia, congestive heart failure, any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or history of myocardial infarction within 6 months prior to first dose with study drug.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as; malabsorption syndrome, resection of the small bowel, or poorly controlled inflammatory bowel disease affecting the small intestine.
* Child-Pugh B cirrhosis (or worse) or a history of hepatic encephalopathy
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
* Patients who need anticancer chemotherapy other than the study drugs during the study or within 4 weeks of study enrollment. Anti-cancer therapy is defined as any agent or combination of agents with clinically proven anti-tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints.
* Patients who need hormonal therapy during the study or within 2 weeks of first study enrollment.
* Patients who need radiotherapy to target lesions during study or within 2 weeks of enrollment.
* Patients who had bone marrow transplant or stem cell rescue.
* Patients who need investigational drug therapy outside of this trial during or within 4 weeks of first study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dae W Kim, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Kim DW, Kim RD, Jimenez MM, Kim Y, Mehta R. A phase II study of trifluridine/tipiracil in combination with ramucirumab in advanced, refractory gastric, or gastroesophageal junction adenocarcinomas. Oncologist. 2025 Dec 1;30(12):oyaf303. doi: 10.1093/oncolo/oyaf303. PMID 41335458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS 102 and Ramucirumab
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAS 102 and Ramucirumab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival defined as the time from starting on trial to date of death from any cause.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS 102 and Ramucirumab
Number analyzed (Participants) | 23
months | 4.8 [4.0 to NA] — Upper limit was not reached

2. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Number of participants with at least one adverse event.
Time Frame: 4 weeks after end of study participation, an average of 6.5 months
Measure: Number; unit: participants
Arm/Group | TAS 102 and Ramucirumab
Number analyzed (Participants) | 23
participants | 23

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, defined as the duration of time from start of treatment to time of progression or death, whichever comes first. Progression is evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS 102 and Ramucirumab
Number analyzed (Participants) | 23
months | 4.9 [4.0 to NA] — Not Reached

4. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate is defined as complete response (CR) + partial response (PR) using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Complete Response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 12 months
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS 102 and Ramucirumab
Number analyzed (Participants) | 18
percentage of participants | 11 [9.622 to 12.578]

ADVERSE EVENTS:
Time Frame: Adverse events collected from first on treatment date to 4 weeks after end of treatment, an average of 6.5 months.
Arm/Group | TAS 102 and Ramucirumab
All-Cause Mortality (participants affected / at risk) | 20/23
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS 102 and Ramucirumab (N=23)
Death NOS (General disorders) | 3 (3)
Sudden death NOS (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Infections and infestations- Other (Infections and infestations) | 1 (1) — Diabetic foot infection
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (3)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS 102 and Ramucirumab (N=23)
Diarrhea (Gastrointestinal disorders) | 13 (15)
Nausea (Gastrointestinal disorders) | 13 (15)
Vomiting (Gastrointestinal disorders) | 12 (15)
Constipation (Gastrointestinal disorders) | 6 (6)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (9)
Toothache (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 14 (16)
General disorders and administration site conditions - Other (General disorders) | 5 (7)
Chills (General disorders) | 4 (5)
Pain (General disorders) | 4 (4)
Edema limbs (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (5)
Flu like symptoms (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (16)
Dizziness (Nervous system disorders) | 6 (6)
Nervous system disorders - Other (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 6 (11)
White blood cell decreased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (4)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (3)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Reproductive system and breast disorders - Other, (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03686488/Prot_SAP_000.pdf